CLINICAL TRIAL: NCT00898703
Title: QUANTIFICATION OF CIRCULATING ENDOTHELIAL CELLS (CEC) AND PLASMA ANGIOGENIC FACTORS IN PATIENTS WITH BREAST CANCER
Brief Title: Studying Blood Samples in Women With Breast Cancer or a History of Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000597587; P30CA023074 (NIH); UARIZ-HSCA01134
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Flow Cytometry; Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: flow cytometry
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with current or previous cancer may help doctors learn more about biomarkers related to cancer.

PURPOSE: This research study is looking at blood samples in women with breast cancer or a history of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare peripheral blood (PB) concentrations of circulating endothelial cells (CEC) in women with measurable, active breast cancer to PB concentrations of CEC in a control population of women with a history of breast cancer who are currently without evidence of active disease.

Secondary

* To compare in women with measurable breast cancer the relationship between PB concentrations of CEC prior to and at 3 and 6 weeks following initiation of a new chemotherapy or hormonal therapy, and correlate these values with clinical response to treatment to determine if CEC can be used as a tumor marker or indicator of disease burden.
* To compare PB concentrations of CEC to levels of plasma proteins associated with angiogenesis, including vascular endothelial growth factor, in women with active or a prior history of breast cancer.

OUTLINE: Peripheral blood and plasma samples are collected for analysis of circulating endothelial cells (CEC) and angiogenic growth factor levels. Blood samples from patients initiating a new chemotherapy or hormonal therapy for breast cancer are collected at baseline and at 3 and 6 weeks following the start of treatment. CEC are quantified via flow cytometry and plasma angiogenic markers are assessed via ELISA.

PROJECTED ACCRUAL: A total of 100 patients with active, measurable breast cancer and 100 patients with a prior history of breast cancer will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Receiving treatment for measurable breast cancer at the Arizona Cancer Center Clinic
  * Being followed for a prior history of breast cancer (with no evidence of active disease) at the Arizona Cancer Center
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women with breast cancer or a history of breast cancer
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2001-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Comparison of levels of peripheral blood (PB) circulating endothelial cells (CEC) and plasma angiogenic factors between patients with active, measurable breast cancer vs prior history of breast cancer with no evidence of active disease

SECONDARY OUTCOMES:
Correlation of CEC and plasma angiogenic factors with response to tumor to a chemotherapy regimen

CONTACTS AND LOCATIONS:
Overall Officials: Alison T. Stopeck, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States